CLINICAL TRIAL: NCT04897685
Title: The Effects of Nature-based Intervention in the Treatment of Depression: Multi-center, Randomized Controlled Trial in Finland
Brief Title: Nature-based Treatment Group for Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: JAMK University Of Applied Sciences (Other)
Collaborators: Tampere University (Other); University of Jyvaskyla (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JAMKUAS
Record Dates: First submitted 2021-05-18; First posted 2021-05-21 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Depression
Keywords: nature-based; therapy group; recovery experiences; nature experiences
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nature-based treatment group (Experimental): The participants in the treatment group were offered 12 nature-based group therapy sessions in addition to standard care.
  Interventions: Behavioral: Flow with Nature
- Control group (No Intervention): The participants in the control group continued treatment as usual in the health care services.

INTERVENTIONS:
Behavioral: Flow with Nature — Nature-based intervention was facilitated by a health care professional and included 12 x 90 mins sessions within 12 weeks.
  Arms: Nature-based treatment group

SUMMARY:
This multi-centre research investigates the effects of nature-based treatment group on participants diagnosed with depression. In total, 147 persons participated in the study in various locations in Finland. All participants received treatment as usual (TAU). They were randomised into nature-based group + TAU (n = 70) or TAU-only (n = 77). The participants in the nature-based group + TAU were offered 12 sessions once a week in addition to standard care. The measurement points included pre-treatment measurement at the baseline and post-treatment measurement at the end of the intervention, which was 12 weeks after the pre-treatment measurement. The follow-up measurement was 3 months after the post-treatment measurement. The effects of the intervention were assessed with a clinical measure of depression (BDI-I) and with indicators of psychological distress (CORE-10), subjective well-being (SWEMWBS), work/study ability (WAI) and nature experiences (ROS, KOLU). The participants in the treatment group (nature-based group +TAU) were compared to the participants in the control group who received TAU-only.

DETAILED DESCRIPTION:
This research investigates the outcomes of nature-based treatment groups in the treatment of adults with depression. In total, 147 participants were involved. Of them, 70 were randomized into DMT group and 77 into the control group. All participants received treatment as usual during the research. The inclusion criteria of the study were: a diagnoses of depression (ICD -diagnostic system), BDI-I score 10 or above (cut off score for mild depression), treatment contact in a health care service and 18-65 years of age. The exclusion criteria were: 1) active suicidal ideation, 2) psychotic symptoms, and 3) substance misuse that is on a critical level (Audit questionnaire scores above 10). Also, participants who had pain-related problems that restricted daily life or were pregnant were not admitted to the study.

Nature-based treatment group was facilitated by a health care professional and included 12 x 90 mins sessions within 12 weeks. Depressive symptoms (BDI-I), psychological distress (CORE-10), subjective well-being (SWEMWBS), ability to work/study (WAI), and nature experiences (ROS, KOLU) were assessed at three measurement points: pre-measurement at the baseline, post-measurement 12 weeks after the pre-treatment measurement, and a follow-up measurement three months after the post-treatment measurement.

This research includes a larger number of participants (N = 147) than have been involved in previous studies utilising randomised controlled trials in nature-based interventions. The research generates further information about the effectiveness of nature-based therapy groups in the rehabilitation of depression as it was conducted in five cities across Finland. This type of multi-centre research can provide a realistic picture of the typical practice of a range of health care professionals working with participants in various geographic locations.

ELIGIBILITY:
Inclusion Criteria:

* A diagnoses of depression (ICD -diagnostic system)
* BDI-I score 10 or above
* Treatment contact in a health care service
* Motivated to commit to a 12-session treatment group taking place in nearby nature environments
* Able to communicate adequately in Finnish in order to participate

Exclusion Criteria:

* Active suicidal ideation
* Psychotic symptoms
* Substance misuse that is on a critical level
* Volunteers who had pain-related problems that restricted daily life or were pregnant were not admitted to the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline depressive symptoms (Beck Depression Inventory; BDI-I) at 12-week post-treatment measurement. | 12 weeks
  BDI-I (Beck Depression Inventory - I) measures depressive symptoms with 21 items. Each item is scored 0-3 and sum scores are calculated on the basis of participants' responses. The total sum score can range from 0 to 63 and higher score indicates higher depression.
Change from post-treatment depressive symptoms (Beck Depression Inventory-I; BDI-I) at three-month follow-up measurement. | 3 months
  The change in depressive symptoms between the post-treatment measurement at the end of the 12-week intervention and the 3-month follow-up. BDI-I (Beck Depression Inventory - I) measures depressive symptoms with 21 items. Each item is scored 0-3 and sum scores are calculated on the basis of participants' responses. The total sum score can range from 0 to 63 and higher score indicates higher depression.

CONTACTS AND LOCATIONS:
Overall Officials: Kalevi Korpela, Professor, Principal Investigator — Tampere University
Locations (3):
- Finland (3):
  - University of Jyväskylä, Jyväskylä
  - Institute of Rehabilitation, JAMK University of Applied Sciences, Jyväskylä
  - Tampere University, Tampere

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Description of the research group — https://research.tuni.fi/enviwell/